CLINICAL TRIAL: NCT03731897
Title: to Evaluate the Efficacy of Prolotherapy Treatment and Compare the Control Group in Patients With Plantar Fasciitis: a Randomized Double-blind Study
Brief Title: Evaluation of the Efficacy of Prolotherapy Treatment in Patients With Plantar Fasciitis: a Randomized Double-blind Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Basak Mansiz-Kaplan, Department of Physical Medicine and Rehabilitation, Ankara Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E171615
Record Dates: First submitted 2018-11-04; First posted 2018-11-06 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2019-07

CONDITIONS: Plantar Fascitis
MeSH Terms: interventions — Glucose; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- prolotherapy (Experimental): Experimental: Plantar fasciitis injection with prolotherapy total 5cc. Procedure: Plantar fascia will be injected to the places where it adheres to the bone.
  Drug: 5 cc 30% dextrose + 4 cc salin + 1cc 2% lidocaine. This treatment, known as regenerative injection therapy, stimulates tissue repair and reduces pain.
  Interventions: Other: 5 cc 30% dextrose + 4 cc salin + 1cc 2% lidocaine.
- control (Placebo Comparator): Placebo Comparator: Plantar fasciitis injection with 9cc salin + 1 cc 2% lidocaine total 5cc.
  Procedure: Plantar fascia will be injected to the places where it adheres to the bone.
  Drug: 9 cc salin + 1cc 2% lidocaine. This treatment is safe for Plantar fasciitis injection.
  Interventions: Other: 9 cc salin + 1cc 2% lidocaine.

INTERVENTIONS:
Other: 5 cc 30% dextrose + 4 cc salin + 1cc 2% lidocaine. — Plantar fascia will be injected to the places where it adheres to the bone.
  Arms: prolotherapy
Other: 9 cc salin + 1cc 2% lidocaine. — Plantar fascia will be injected to the places where it adheres to the bone.
  Arms: control

SUMMARY:
Plantar fasciitis is the most common cause of heel pain and it is diagnosed by clinically.

Resting, stretching exercises, weight loss, nonsteroidal anti-inflammatory drugs and physical therapy methods are used in the treatment. Steroid injection can be applied in patients who do not respond to these treatments. But steroid injection is not a pathology-based treatment, and also can cause serious side effects, such as fat pad atrophy and plantar fascia rupture. At this stage, in patients who do not respond to conservative treatments, new methods such as dextrose prolotherapy and platelet rich plasma may be used instead of steroid injection. In the literature, there is insufficient study showing effect of prolotherapy in patients with plantar fasciitis. Because these studies enrolled small number of patients and lacked controlled design. The investigators design a randomized, double-blind, controlled trial to assess the effect after prolotherapy injection in patients with plantar fasciitis.

The participants evaluated with clinically and sonographically. The aim of this study is to compare the pain, function and thickness of proximal plantar fascia in prolotherapy or control group.

DETAILED DESCRIPTION:
After obtaining written informed consent, patients of clinically and sonographically diagnosed with plantar fasciitis were randomized into intervention and control group. Participants in intervention group received two-session prolotherapy injection and control group received two-session 9cc salin + 1 cc 2% lidocaine injection in 3 weeks interval. Stretching and range of motion exercises were prescribed after treatment.

The primary outcome is visual analog scale (VAS) and secondary outcomes include Foot Function Index , ultrasonographic measurement of proximal plantar fascia. The evaluation was performed pretreatment as well as on the 1st and 3th month the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-65 year-old.
* Heel pain for at least 3 months
* Plantar fasciitis which diagnosed clinically and confirmed using ultrasonography (plantar fascia thickness > 4mm)

Exclusion Criteria:

* History of chronic pain syndromes
* Patients undergoing steroid injections for the treatment of plantar fasciitis in the last 6 months
* Rheumatic diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-11-12 (Actual); Primary Completion 2019-03-12 (Actual); Study Completion 2019-06-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline of pain on 1st and 3th months after treatment: VAS | Pre-treatment, 1st and 3th months after treatment
  Using the Visual analog scale (VAS) to measure the pain scale before treatment and multiple time frame after treatment. Recorded on a visual analogue scale (VAS), scores range from 0 to 100 mm, with higher scores indicating worse pain.

SECONDARY OUTCOMES:
Change from baseline in activity and functional status on 1st and 3th months after treatment. | Pre-treatment, 1st and 3th months after treatment
  Using the Foot Function Index (FFI) to measure the activity and functional status before treatment and multiple time frame after treatment. . The FFI consists of 23 self-reported items divided into 3 subcategories on the basis of patient values: pain, disability and activity limitation. The patient has to score each question on a scale from 0 (no pain or difficulty) to 10 (worst pain imaginable or so difficult it requires help), that best describes their foot over the past week. The higher scores indicate worse pain. Both total and subcategory scores are calculated.
Change from baseline in thickness of proximal plantar fascia on 1st and 3th months after treatment. | Pre-treatment, 1st and 3th months after treatment treatment
  Using the musculoskeletal sonogram to measure the proximal plantar fascia thickness.

CONTACTS AND LOCATIONS:
Overall Officials: Basak Mansiz-Kaplan, Principal Investigator — Physical Medicine and Rehabilitation
Locations (1):
- Basak Mansiz-Kaplan, Ankara, Turkey (Türkiye)